CLINICAL TRIAL: NCT04204083
Title: A Prospective Study of a Single Injection Cross-linked Sodium Hyaluronate (MONOVISC) to Provide Symptomatic Relief of Osteoarthritis of Hip Joint
Brief Title: MONOVISC for Hip Joint Pain Relief Due to Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anika Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MON 18-01
Record Dates: First submitted 2019-12-17; First posted 2019-12-18 (Actual); Results first posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Osteoarthritis, Hip
Keywords: Hyaluronic acid
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Monovisc (Experimental): Single injection of Monovisc into the index hip joint
  Interventions: Device: Monovisc

INTERVENTIONS:
Device: Monovisc — A chemically cross-linked sodium hyaluronate supplied as a 4 mL unit dose in a 5 mL glass syringe.

SUMMARY:
Obtain real world, post market data to confirm the clinical improvement and safety in patients treated with a single injection of MONOVISC for the symptomatic relief of osteoarthritis in the hip joint.

DETAILED DESCRIPTION:
This is a prospective, post market clinical follow-up (PMCF) multi-center, open-label study to evaluate the residual risk of injections of MONOVISC for relief of pain in patients with a diagnosis of an osteoarthritic hip joint.

The subjects in this study will be patients with a diagnosis of osteoarthritic (OA) joint who the investigator determines are appropriate candidates for treatment with a viscoelastic injection of MONOVISC.

Up to 25 subjects will be enrolled at up to 20 investigational sites in the EU. Subject participation will last approximately 6 Months, with visits scheduled at Screening, Baseline, 1 month, 3 month and 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Body Mass Index (BMI) ≤ 35 kg/m2
3. Diagnosis of symptomatic osteoarthritic joint in the index joint (Kellgren-Lawrence grade I to III) to be treated with MONOVISC injection.
4. Failed conservative treatment for joint osteoarthritis.
5. NRS pain on walking ≥4 and ≤ 9 in index joint.
6. Subject must be willing to abstain from other treatments of the index joint for the duration of the study.
7. Subject is willing to discontinue all analgesics including NSAIDs, except acetaminophen/paracetamol, at least seven days before the treatment injection and through the completion of the study.
8. Subject is willing to use only acetaminophen/paracetamol (up to a maximum of 4.0 grams per day per the package insert) for the treatment of joint pain for the duration of the study. At least forty-eight hours prior to the Baseline Visit and each follow-up visit, the subject is willing to discontinue use of acetaminophen/paracetamol.
9. Subject is willing to maintain a stable dose of oral glucosamine and/or chondroitin sulfate products throughout the study, if taken prior to signing the informed consent form (ICF).
10. Able and willing to provide signed informed consent.

Exclusion Criteria:

1. History of hypersensitivity to any of the ingredients in the hyaluronan
2. Infection or skin disease in the area of the injection site or index joint
3. NRS pain on walking > 3 in the contralateral joint
4. NRS pain on walking > 3 in the ipsilateral knee or ankle
5. Subject received an injection of Hyaluronic Acid (HA) and/or steroid in either joint within 6 months of signing the informed consent form (ICF). A subject will be excluded if they are planning to receive an HA or steroid injection (other than the study injection) in either joint during the course of this study.
6. Known inflammatory or autoimmune disorders (including rheumatoid arthritis, gout), or other pre-existing medical conditions that, in the opinion of the investigator, could impact treatment of the index joint or affect the ability of the subject to accurately complete the study questionnaires and comply with the study requirements.
7. Subject is taking medications at the time of signing the ICF which could interfere with the treatment procedure, healing and/or assessments. This includes but is not limited to oral or injectable anticoagulant treatments, anti-aggregant platelet treatment, chronic opioid analgesics. Low dose aspirin used for cardiovascular protection is allowed if a stable regimen is maintained for the duration of the study.
8. Subjects who had an oral, intramuscular, intravenous, rectal suppository or topical (excluded in index joint only) corticosteroid prior 30 days of signing the ICF are excluded. Topical corticosteroid use at any site other than the index joint is allowed.
9. Significant trauma to the index hip within 26 weeks of screening
10. Chronic use of narcotics or cannabis.
11. Ligament instability or tear in index joint.
12. Diagnosis of fibromyalgia
13. Diagnosis of osteonecrosis in index joint
14. Subject has significant varus or valgus deformity greater than 10 degrees in either knee.
15. Subject requires consistent use of an assistive device (e.g. wheelchair, walker, etc.) Occasional use of a cane is acceptable.
16. Uncontrolled diabetes with HbA1c of >7%.
17. Subject is a woman who is pregnant or breastfeeding at the Screening Visit or a woman of child bearing potential who refuses to use effective contraception during the course of the study.
18. Subject is receiving or in litigation for worker's compensation.
19. Otherwise determined by the investigator to be medically unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kara Mezger, Study Director — Anika Therapeutics
Locations (4):
- Krajská zdravotní, a.s., Ústí nad Labem, Czechia
- Poland (3):
  - Nzoz Medi-Spatz, Gliwice
  - SPORTO, Lodz
  - Przychodnia Rodzinna na Sadowej, Torun

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only one hip [Index Hip] of each participant was included in this study
Period: Overall Study
Arm/Group | Monovisc
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Monovisc
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.72 (10.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0
Index Hip [Count of Participants; unit: Participants]
  Right | 13
  Left | 12

OUTCOME MEASURES:

1. Primary Outcome: Numerical Rating Scale (NRS) Pain on Walking
Description: Mean Change in Numerical Rating Scale (NRS) Pain on Walking in the Index Hip from baseline to 6 Months post injection. NRS is an 11-Point scale where 0=No Pain, 10=Worst Pain. A larger negative value (maximum -10.0) for the change from baseline indicates less pain and a better outcome following treatment.
Time Frame: From Baseline to 6 Months
Population: Intent To Treat (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Monovisc
Number analyzed (Participants) | 25
score on a scale | -3.68 (2.87)
Statistical Analysis 1: Comparison: Monovisc; Test type: Other; p < 0.0001, t-test, 1 sided — P-Value was calculated

2. Secondary Outcome: Lequesne Hip Index Score
Description: Mean change in Lequesne Hip Index Score from baseline to 6 months post injection. The Lequesne Hip Index is a three-section patient questionnaire that evaluates (1) pain or discomfort, (2) maximum distance walked, and (3) activities of daily living with 0 = best results / normal scores, to scores >14 = extremely severe, to a maximum index score of 24 points.
  A negative value for the change in Lequesne Hip Index indicates improvement. A larger negative value indicates a higher level of improvement, and a better outcome.
Time Frame: From Baseline to 6 Months
Population: Intent To Treat (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Monovisc
Number analyzed (Participants) | 25
score on a scale | -5.20 (3.46)
Statistical Analysis 1: Comparison: Monovisc; Test type: Other; p < 0.0001, t-test, 1 sided — P-Value was calculated

3. Secondary Outcome: Patient Global Assessment (PGA)
Description: The change from baseline to 6 months in hip pain post-treatment as measured by the Patient Global Assessment (PGA) Score. PGA Score records participant responses to their assessment of how much their STUDY (treated) hip is bothering them today . The PGA Score is a validated 11-point Likert scale ranged from 0 = No Pain to 10 = Worst Pain.
  A negative value for the change from baseline indicates improvement in PGA Score. A larger negative value indicates less pain, and a better clinical outcome.
Time Frame: From Baseline to 6 Months
Population: Intent To Treat (ITT)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Monovisc
Number analyzed (Participants) | 25
score on a scale | -3.52 (3.14)
Statistical Analysis 1: Comparison: Monovisc; Test type: Other; p < 0.0001, t-test, 1 sided — P-Value was calculated

4. Secondary Outcome: The Outcomes Measures for Rheumatic Arthritis Clinical Trials-Osteoarthritis Research Society International (OMERACT-OARSI) Responder Index
Description: The post-treatment responder rate at 6 months is determined through a calculation defined by the Outcomes Measures for Rheumatic Arthritis Clinical Trials-Osteoarthritis Research Society International (OMERACT-OARSI) Responder Index. The OMERACT-OARSI Responder Index reports the percentage of subjects that met the criteria to be a good responder to treatment. The criteria for response are (1) improvement in pain or physical function >50% and an absolute change >20 mm; or (2) improvement of >20% with an absolute change >10 mm in at least of the following three categories: pain, physical function, and patient's global assessment.
  A higher percentage of subjects responding indicates a better clinical outcome.
Time Frame: 6 Months
Population: Intent To Treat (ITT)
Measure: Count of Participants; unit: Participants
Arm/Group | Monovisc
Number analyzed (Participants) | 25
Participants | 20

5. Secondary Outcome: Number of Participants NOT Using Rescue Medication (Acetaminophen/Paracetamol)
Description: The usage of Rescue Medication (RM) as based on the number of participants at 6 months post treatment that were NOT using acetominophen/paracetamol RM for pain or discomfort.
  A larger percentage of participants that were NOT using RM may correlate to a better clinical outcome in terms of pain.
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Monovisc
Number analyzed (Participants) | 25
Participants | 21

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from the time of the Baseline Study Visit until Study Completion at 26 Weeks (6 months).
Description: The definitions of adverse events and serious adverse events is the same as used in the clinicaltrials.gov definitions.
  The incidence, timing, severity, and relationship to treatment of all Adverse Events (AE) were collected and coded using Medical Dictionary for Regulatory Activities (MedDRA).
Arm/Group | Monovisc
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 9/25
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Monovisc (N=25)
Viral pharyngitis (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Oral herpes (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Diabetes insipidus (Endocrine disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
There were no limitations or caveats associated with the conduct of this trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
INVESTIGATOR may publish the Data/Results with the consent of the SPONSOR if:

1. Publication is done after primary publication covering data from all participating sites, and provided the Data/Results do not contain any Confidential Information.
2. Eighteen (18) months has elapsed after entire completion of the Clinical Trial at all participating sites.

DOCUMENTS (2):
  • Study Protocol (2019-07-11): https://cdn.clinicaltrials.gov/large-docs/83/NCT04204083/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-09): https://cdn.clinicaltrials.gov/large-docs/83/NCT04204083/SAP_001.pdf